CLINICAL TRIAL: NCT06465615
Title: Effect of Binocular Dichoptic Reading Treatment on Visual Function in Children With Symptomatic Convergence Insufficiency: a Pilot Noninferiority Study. ALEDICE
Brief Title: Effect of Binocular Treatment Using a Dichoptic Reading Application in Children With Convergence Insufficiency.
Acronym: ALEDICE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL22_0552
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-05

CONDITIONS: Ophthalmological Disorder
Keywords: Convergence insufficiency; therapy, Vision, Binocular; physiology, Vision, Monocular; physiology, Depth Perception; physiology, Contrast Sensitivity
MeSH Terms: conditions — Eye Diseases; Ocular Motility Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized, controlled, non-inferiority, open-label study with blinded assessment of primary endpoint.
Who Masked: Care Provider
Masking Description: An orthoptist fwho may also be in charge of rehabilitation, will carry out the initial assessment (near convergence amplitude, punctum proximum of convergence,...).
  Another orthoptist will perform the same assessments at S3 and S6, blinded to the treatment arms and initial measurements to avoid bias:
  Another orthoptist in the department, different from the blinded orthoptist, will provide conventional rehabilitation and will not be blinded to the treatment groups assigned to his or her patients. This orthoptist designated for rehabilitation may also be in charge of the initial evaluation.
  The department's CRA will be vigilant from the outset to define who will be the blinded orthoptist assessor (assessments at S3 and S6) and the orthoptist rehabilitator and/or assessor for the initial visit. Randomization will be carried out by a CRA, who will only reveal the randomization arm to the orthoptist designated for rehabilitation and/or initial assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): self-rehabilitation at home. Intervention 25 min/day, 5 days a week for 6 weeks at home (weekly load of 125 minutes), on a dichoptic reading application on a loaned digital tablet, wearing anaglyph glasses provided and patient's optical correction (if applicable).
  Interventions: Device: Self-education with dichoptic reading on tablet
- Control group (Active Comparator): The control group will receive conventional treatment consisting of 12 sessions of 25 minutes each over 6 weeks of rehabilitation with an orthoptist in the ophthalmology department of Montpellier University Hospital.
  Interventions: Procedure: Conventional orthoptic rehabilitation

INTERVENTIONS:
Device: Self-education with dichoptic reading on tablet — Intervention 25 min/day, 5 days a week for 6 weeks at home (125-minute weekly load), under the supervision of a parent, on a dichoptic reading application on a loaned digital tablet, wearing anaglyph glasses provided and the patient's optical correction (if applicable).
  During the first half of treatment (first 3 weeks), dichoptic separation takes place at the word level, and during the second half of treatment (last 3 weeks), it takes place at the individual letter level to promote precise eye alignment. This shift from dichoptic separation at word level to letter level increases the difficulty of the task. The text is freely chosen by the child and parent from a bank of age-appropriate books.
  Arms: Experimental group
Procedure: Conventional orthoptic rehabilitation — Conventional orthoptic rehabilitation consisting of 12 x 25-minute sessions twice a week over 6 weeks, carried out with an orthoptist from Montpellier University Hospital, combined with reinforcement exercises to be carried out at home for 15 minutes a day under parental supervision, 5 days a week (125-minute weekly load). This is the standard orthoptic treatment offered in France to patients with symptomatic convergence insufficiency, according to orthoptic procedures (10-15 sessions of the order of 20-25 minutes and 10-15 minutes of daily reinforcement exercises at home).
  Arms: Control group

SUMMARY:
Convergence insufficiency is a common disorder of binocular vision that can appear as early as childhood after visual effort, and is often associated with a variety of symptoms such as eyestrain, headaches, blurred vision and diplopia.

Treatment of symptomatic convergence insufficiency generally involves the intentional and controlled manipulation of a visual target's blur, conjugate and vergence movements around this target, with the aim of normalizing the accommodation and vergence systems and their mutual interactions.

Despite the effectiveness of this treatment, compliance is not optimal, ranging from 24% to 91% in the youngest patients. One of the main challenges is to keep patients focused and interested during the potentially tedious and repetitive periods of over-convergence. In order to stimulate the patient's active participation and stable, sustained attention, a dichoptic reading application on a digital tablet has been developed to provide sustained training in ocular alignment and coordination to reduce symptoms and restore binocular function in patients with symptomatic convergence insufficiency.

DETAILED DESCRIPTION:
The dichoptic reading application on a digital tablet consists in reading, with red-green anaglyph glasses, a text composed of letters or words presented both binocularly and monocularly (black and red-green, respectively) from downloaded e-books. After centralized randomization, patients will undergo either reference orthoptic rehabilitation (control group) or dichoptic treatment on a digital tablet (experimental group). The control group will receive 12 training sessions (25 minutes twice a week for 6 weeks) as part of their regular treatment in the Ophthalmology Department of the CHU de Montpellier, while the experimental group will perform self-training at home (25 min/day, 5 days a week for 6 weeks). For all participants, an initial visit and two follow-up evaluation visits (visits 2 and 3) will be scheduled 3 and 6 weeks (+ 1 week) after the start of the intervention, and will be carried out by one of the 3 other orthoptists in the Ophthalmology Department of the CHU de Montpellier.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8 to 17
* Minimum current schooling: CE2 class
* Availability of at least one legal guardian to supervise the child's training (strengthening exercises to be performed at home 15 min/day for the control group/ 25 min/day session at home for the experimental group) and complete the patient logbook.
* Ophthalmological check-up performed within 2 months prior to inclusion
* Convergence Insufficiency Symptom Survey (CISS) score ≥ 16
* Convergence punctum proximum ≥ 6 cm
* Amplitude of fusion in near convergence ≤ 15 prismatic dioptres or less than 2 times the phoria measured in near vision (Sheard's criterion).
* Best corrected distance and near visual acuity ≥ 20/25 (=8/10) and wearing appropriate refractive correction (glasses or contact lenses) for at least 2 weeks prior to study inclusion.
* See letters/words and be able to read 3 complete sentences on a predefined text presented dichoptically on the tablet with anaglyph glasses
* Availability of the patient to complete the training protocol over 6 weeks (or a maximum of 9 weeks in the event of temporary interruption of treatment).

Exclusion Criteria:

* Binocular vergence dysfunctions such as constant strabismus
* Prism (unless removed ≥ 2 weeks prior to inclusion)
* History of recent orthoptic rehabilitation (< 6 months)
* History of intraocular or refractive surgery
* Current amblyopia treatment or treated amblyopia (isoacuity) < 6 months
* Best corrected visual acuity of the worse eye < 8/10
* Medication that may interfere with binocular vision and/or accommodation
* Accommodation paralysis
* Ocular comorbidity likely to reduce visual acuity
* History of vestibular migraines, vestibular disorders
* History of ocular or systemic disease, infections/congenital malformations
* Neurological history: stroke, head trauma, tumors, epilepsy or neurodegenerative disorders
* Specific learning disability
* Developmental delay (global, language, learning) likely to interfere with treatment or evaluation.
* Failure to obtain written informed consent after a period of reflection
* Not being affiliated to a French social security scheme or benefiting from such a scheme
* Pregnant or breast-feeding

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of symptoms at the end of the intervention | T0 and T6 weeks
  Evolution of symptoms assessed via the Convergence Insufficiency Symptom Survey (CISS) score, version 15, measured before and 6 weeks after the start of the intervention in children with convergence insufficiency.
Evolution of symptoms halfway through the intervention | T0 and T3 weeks
  Evolution of symptoms (decrease in Convergence Insufficiency Symptom Survey (CISS) score measured 3 weeks after the start of binocular treatment)

SECONDARY OUTCOMES:
Evolution of the punctum proximum of convergence (PPC) | T0 and T3 weeks and T0 and T6 weeks
  This test defines the closest point of fixation to the patient on which the 2 eyes can converge and see simply. It is measured using the Astron ACR/21 international accommodative rule.
Evolution of stereoacuity | T0 and T3 weeks and T0 and T6 weeks
  The McGill clinical stereo test (McGill University) evaluates relief vision (threshold expressed in arcseconds) through a digital tablet with red-green anaglyph glasses.
Normalization of fusion amplitude in near convergence | T0 and T3 weeks ans T0 and T6 weeks
  A fusion amplitude in near-normal convergence is defined as greater than 15Δ and satisfying Sheard's criterion.
Normalization of punctum proximum of convergence (PPC) | T0 and T3 weeks ans T0 and T6 weeks
  A normal convergence punctum proximum is defined as less than 6 cm.
Evolution of reading speed | T0 and T3 weeks ans T0 and T6 weeks
  reading speed assessed by the Minnesota Low Vision Reading Test (MNREAD) in seconds.
Interocular suppression measured with the Dichoptic Contrast Ordering Test (DICOT) | T0 and T3 weeks ans T0 and T6 weeks
  Interocular suppression measured with the Dichoptic Contrast Ordering Test (DICOT)
Changes in quality of life | T0 and T3 weeks ans T0 and T6 weeks
  Quality of life measured with the Pediatric Quality of Life Inventory (PedsQL)
Prevalence of patients with "Complete Response", "Partial Response" and "Nonresponders | T3 weeks and T6 weeks
  Prevalence of patients with "Complete Response", "Partial Response" and "Nonresponders", defined as follows:
  Complete response :
  * ISSC score <16
  * AND normal convergence punctum proximum (i.e. less than 6 cm)
  * AND normal near convergence fusion amplitude (i.e. greater than 15Δ and satisfying Sheard's criterion).
  Partial response:
  * CISS score <16 or 10-point decrease in CISS
  * AND :
    * Normal convergence punctum proximum
    * OR improvement in convergence proximal punctum of more than 4 cm
    * OR normal near convergence fusion amplitude
    * OR increase in near convergence fusion amplitude by more than 10Δ. Non-responders: Patients not meeting the criteria for success or improvement.
Treatment compliance | T3 weeks and T6 weeks
  For the experimental group, compliance is measured using a percentage of training sessions completed, obtained from automatic recording by the tablet software and the patient diary, in which the date and duration (seconds) of each training session are recorded. For the control group, compliance is measured using a percentage combining the number of training sessions performed (collected by the orthoptist) and home exercises (self-reported by the patient), with dates and durations recorded in a patient logbook.
Adherence to self-training | T3 weeks and T6 weeks
  Adherence to self-training evaluated in a patient logbook: training time completed vs. training time planned.
Visual comfort when using the dichoptic reading application | T3 weeks and T6 weeks
  Measurement of visual comfort when using the dichoptic reading application with the modified Convergence Insufficiency Symptom Survey score.The modified Convergence Insufficiency Symptom Survey score ranges from 0 to 60. Higher scores mean a worse outcome, indicating a high presence of symptoms.
Level of certainty of recognition of the patient randomization arm for the evaluating orthoptist | T3 weeks and T6 weeks
  Likert scale assessing the evaluator's level of certainty regarding recognition of the patient's allocation to the experimental arm. The modified Convergence Insufficiency Symptom Survey score ranges from 0 to 4. higher scores mean a better outcome, indicating a low level of certainty of recognition of patient randomization arm.
Adverse events | T3 weeks ands T6 weeks
  Collection of adverse events self-reported by the patient and collected by the medical team during assessment visits.

IPD SHARING:
Plan to Share IPD: No